CLINICAL TRIAL: NCT00410111
Title: A Pilotstudy on Pathogenesis and Cerebrovascular Manifestations of Septic Encephalopathy
Brief Title: Pathogenesis and Cerebrovascular Manifestations of Septic Encephalopathy
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Other Study IDs: EKBB 226/06
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Sepsis
Keywords: sepsis; encephalopathy; cerebral perfusion; electroencephalogram
MeSH Terms: conditions — Sepsis; Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Septic encephalopathy is an important complication of sepsis. Why some patients with sepsis develop septic encephalopathy is unknown. We will investigate whether patients who develop this condition have different patterns of cerebrovascular reactivity and whether it is possible to predict the development of septic encephalopathy from early measurements of cerebral perfusion or from the EEG. We will specifically test the hypotheses that septic encephalopathy may not be predicted by changes in the EEG, and that cerebrovascular autoregulation is not dysfunctional in septic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis
* Admission to ICU

Exclusion Criteria:

* CNS infection
* History of cerebrovascular disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with sepsis, severe sepsis or septic shock admitted to an intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2007-01; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luzius A Steiner, MD PhD, Principal Investigator — Department of Anesthesia, University of Basel Hospital, Basel, Switzerland
Locations (1):
- Operative Intensivbehandlung, University of Basel Hospital, Basel, Switzerland

REFERENCES:
- [Derived] Pfister D, Siegemund M, Dell-Kuster S, Smielewski P, Ruegg S, Strebel SP, Marsch SC, Pargger H, Steiner LA. Cerebral perfusion in sepsis-associated delirium. Crit Care. 2008;12(3):R63. doi: 10.1186/cc6891. Epub 2008 May 5. PMID 18457586